CLINICAL TRIAL: NCT04884789
Title: Tolerance Assessment of Tailored 3d-printed Transparent Face Orthosis With Silicone Interface for the Treatment of Post-burn Face Scar
Brief Title: Tolerance Assessment of Tailored 3d-printed TFO With Silicone Interface for the Treatment of Post-burn Face Scar
Acronym: ECORCE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal investigator departure
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2018-A03067-48
Record Dates: First submitted 2021-02-25; First posted 2021-05-13 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Burn Scar
Keywords: Burns; Transparent Face Orthosis; Silicone application; 3d Printed; Face
MeSH Terms: conditions — Burns; Facies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Post-Burn Face scar (Experimental): Use of 3d printed TFO with silicone interface (COFIS 3D)
  Interventions: Device: COFIS 3D

INTERVENTIONS:
Device: COFIS 3D — Patient have to wear the COFIS 3D 20h a day for at least 6 month
  Other Names: 3d printed Transparent Face Orthosis with silicone interface

SUMMARY:
The purpose of this study is to assess the tolerance of tailored 3d-printed transparent face orthosis used in the medical care of post-burn face scar.

DETAILED DESCRIPTION:
Burn injuries are not a rare affection. According to WHO (World Health Organization), in 2004 there were 11 million peoples in the world who were affected by burn injuries caused by fire and who needed medical cares. This important number ignores non-fire thermal, chemical and electrical burns. Face is one of the most susceptible areas of burn where the prevalence was reported to be 6-60%.

Hypertrophic scars (HS) are frequent consequences of dermal burn with a prevalence of 70% of burned people. HS, which are a dermal fibro-proliferation, are rigid, erythematous and thickened scars associated with pigmentation abnormalities, xerosis, thermal sensitivity, pain and pruritus.

When HS is located on the face, they can cause cosmetic disorder with disfigurement and psychological distress.

Pressure therapy and silicone application are the two recommended non-invasive care for prevention and treatment of hypertrophic scarring after burn. On the face, Pressure Garment Therapy (PGT) cannot exert the required pressure because of concave or flat shape so the use of face mask is the most common form of pressure therapy on the face.

The face mask manufacturing is artisanal, time consuming and variable between all burn centers. They are not very accurate and have difficulties to apply effective pressure on certain face areas such as nasolabial folds.

Our Transparent Face Orthosis (TFO) uses tri-dimensional cam for measurement and 3d-printing technology for manufacturing. We think this way to manufacture the TFO will be more accurate and efficient, less expansive and time consuming. Moreover, the addition of a silicone interface between the TFO and the face will associate silicone application therapy and pressure therapy what should be more effective than pressure therapy alone.

The purpose of this study is to assess the tolerance of tailored 3d-printed transparent face orthosis used in the medical care of post-burn face scar.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Post-Burn Face scar during maturation stage or surgical intervention on post-burn face scar during maturation stage
* Patient agrees to shave beard if necessary for 3D camera measurement
* Patient able to express informed consent
* Affiliation to a social security scheme

Exclusion Criteria:

* Post burn face scar in the sequela stage
* Patient with unbalanced photosensitive epilepsy
* Patient with an unconsolidated fracture of the face's bones or skull
* Patient with a known allergy to silicone
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Number of Local Side Effects | Month 1
  wound, device related pain, rash, temporomandibular joint pain, dental pain, suffocating sensation

SECONDARY OUTCOMES:
Evaluation of scar evolution with VSS | Month 1; Month 6; Month 12; Month 18; Month 24
  Vancouver Scar Scale (VSS) assesses 4 variables: vascularity (range 0-3), height/thickness (range 0-3), pliability (range 0-5) and pigmentation (0-2). A total scores ranges from 0 to 13, whereby a score of 0 reflects normal skin.
Evaluation of scar evolution with POSAS | Month 1; Month 6; Month 12; Month 18; Month 24
  Evaluation of scar evolution by Patient and Observer Scar Assessment Scale (POSAS). It consists of two scales which assesses vascularity, pigmentation, thickness, relief, pliability, and surface area and it incorporates patient assessment of pain, itching, color, stiffness, thickness and relief. All items were evaluated on numerical rating scales ranging from 1 to 10 (with 10 indicating the worst score).
Wearing time | Month 1; Month 6; Month 12; Month 18; Month 24
  Diurnal and nocturnal wearing time in hours
Manufacturing time | Month 1; Month 6; Month 12; Month 18; Month 24
  Time of device's manufacturing
Reprints | Month 1; Month 6; Month 12; Month18; Month 24
  Number of reprints needed per patient
Device lifetime | Month 1; Month 6; Month 12; Month18; Month 24
  Device lifetime corresponds to the time between implementation and change of device (for any Reason) in days
Evaluation of the quality of life with the BSHS-B | Month 1; Month 6; Month 12; Month 18; Month 24
  Evaluation of the quality of life of patients by the BSHS-B (Burn Specific Health Scale - Brief). The BSHS-B consists of 40 items divided into four domains with nine subscales (heat sensitivity, affect, hand function, treatment regimens, work, sexuality, interpersonal relationships, simple abilities and body change). Items are answered on a 5-point Likert scale ranging from 0 (extremely) to 4 (not at all).
Number of Local side effects | Month 6
  wound, device related pain, rash, temporomandibular joint pain, dental pain, suffocating sensation

CONTACTS AND LOCATIONS:
Overall Officials: Clémence DEFFINIS, MD, Principal Investigator — CHR Metz Thionville